CLINICAL TRIAL: NCT03049553
Title: Trial23 - A Method Study on the Use of Primary HPV-testing With Cytology Triage in Women Offered HPV-vaccination as Girls
Brief Title: Trial23 - A Method Study on Cervical Screening in Women Offered HPV-vaccination as Girls
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Copenhagen (Other)
Collaborators: Naestved Hospital (Other); Aalborg University Hospital (Other); Soenderjylland Hospital (Unknown); Esbjerg Hospital - University Hospital of Southern Denmark (Other); Randers Regional Hospital (Other)
Responsible Party: Principal Investigator, Elsebeth Lynges, Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 102-2793/15-3000
Record Dates: First submitted 2017-01-31; First posted 2017-02-10 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Cervical Intraepithelial Neoplasia (CIN)
Keywords: Cervical screening; Human papillomavirus (HPV); Cytology; HPV-test; Cervical intraepithelial neoplasia (CIN)
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HPV-test (Other): Cobas HPV-DNA test is performed on the cervical sample in addition to the routine cytology
  Interventions: Device: Cobas HPV-DNA test
- Routine (No Intervention): Screening with cytology as usual in the cervical screening program

INTERVENTIONS:
Device: Cobas HPV-DNA test — Cobas HPV-DNA testing device from Roche is already in standard use in the Danish screening program for purpose of triage and primary screening of women 60+. It has four signals; HPV-negative, HPV-16, HPV-18 and "other"
  Arms: HPV-test

SUMMARY:
In Denmark, the first birth cohorts of women offered HPV-vaccination as girls are entering the cervical screening program. These women are expected to be better protected against cervical cancer. It has not yet been decided how to screen these women.

This method study will investigate a possible screening scheme that could provide a reduced burden of screening for HPV-vaccinated birth cohorts.

DETAILED DESCRIPTION:
In Denmark, women aged 23-49 are offered cervical screening with liquid-based cytology (LBC) every 3rd year, and women aged 50-59 every 5th year. Women aged 60-64 are offered an exit HPV-DNA test.

In 2008 vaccination against Human papilloma virus (HPV) was offered free of charge to girls aged 13-15. HPV-vaccination has been part of the child vaccination program for 12-year old girls since 2009. Women born in 1994 were offered HPV-vaccination at age 14, and approximately 80% are HPV-vaccinated. These women entered the screening program in 2017.

HPV-testing is shown to provide a better protection against cervical cancer than cytology testing, and the 6-year protection against CIN3+ after a negative HPV-test has been observed to be higher than the 3-year protection after a negative cytology test (ref).

The aim of the study is to evaluate if primary screening with HPV-testing and LBC triage every 6 years in women offered HPV-vaccination as girls would provide at least the same protection as the present screening, measured by cumulative number of cervical intraepithelial neoplasia (CIN). This screening scheme would allow HPV-negative women to benefit from a prolonged screening interval and thereby reduce the burden of screening for HPV-vaccinated birth cohorts.

The study is deemed a method study by the ethical committee of the Capital region and informed consent is, therefore, not required. The study is approved by the Danish data protection agency.

The study will be undertaken as a method study embedded in the existing cervical screening program in the study area: Region Zealand, Northern Denmark region, Central Denmark region and part of region of Southern Denmark. The study is planned to run over three screening rounds. We expect 12000 women to be screened in the baseline screening round.

The study includes all women born in 1994 who live in the study area and participate in cervical screening. For a random half of these women, an HPV-DNA test is performed in addition to routine cervical cytology. The result of the HPV-test will not affect screening or follow-up, but is performed solely for purposes of the method study. CINtec p16 histology will be performed on all cervical biopsies in the study to ensure the quality of the diagnosis.

When screening samples are received at the pathology labs the allocation (HPV+/- in addition to cytology) will appear automatically in the IT-system.

The study will be conducted a non-inferiority study. If non-inferiority is declared, analysis for superiority will be conducted. Censoring will be performed in the event of death, emigration, end of study and at first cervical intraepithelial neoplasia grade 3 or above (CIN3+) or conization. Data on primary and secondary endpoints will be collected from National Health registers.

The project is supported by funds from 'Det Frie forskningsråd', 'Helsefonden' and 'Johannes Clemmesens Forskningsfond'. Cobas HPV-DNA and CINtec p16 histology test-kits are sponsored by Roche. Both tests were in standard use in the pathology departments prior to the project.

Results of the baseline screening round and final results from the study will be published in relevant peer-reviewed journals.

ELIGIBILITY:
Inclusion Criteria:

* Women born in 1994 living in the study area

Exclusion Criteria:

* None, as it is a public health trial

Ages: 23 Years to 23 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7000 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Cumulative CIN3+ (cervical intraepithelial neoplasia grade 3 and above) in baseline screen-negative women. | After up to 9 years follow-up (end-of-study)
  Histologically proven CIN3+ is chosen as primary outcome measure because it is the diagnostic threshold above which conization is recommended by the Danish Society of Gynecology and Obstetrics. Primary outcome will be based on intention-to-treat and per protocol analysis and stratified by region of residence. Primary HPV-testing with cytology triage every six years compared to cytology every three years will be approximated from the observed data.

SECONDARY OUTCOMES:
Cumulative CIN3+ overall | After up to 9 years follow-up (end-of-study)
  Intention-to-treat and per protocol analysis. Stratified by region of residence.
Cumulative CIN2 (cervical intraepithelial neoplasia grade 2) overall | After up to 9 years follow-up (end-of-study)
  Intention-to-treat and per protocol analysis. Stratified by region of residence.
Cumulative CIN2 in baseline screen-negative women | After up to 9 years follow-up (end-of-study)
  Intention-to-treat and per protocol analysis. Stratified by region of residence
Cumulative CIN1 (cervical intraepithelial neoplasia grade 1) overall | After up to 9 years follow-up (end-of-study)
  Intention-to-treat and per protocol analysis. Stratified by region of residence
Cumulative CIN1 in baseline screen-negative women | After up to 9 years follow-up (end-of-study)
  Intention-to-treat and per protocol analysis. Stratified by region of residence

OTHER OUTCOMES:
Baseline CIN1 | After up to 2 years follow-up
  Number of women with the secondary outcome in the two study arms at baseline (baseline screening round).
Baseline CIN2 | After up to 2 years follow-up
  Number of women with the secondary outcome in the two study arms at baseline (baseline screening round).
Baseline CIN3+ | After up to 2 years follow-up
  Number of women with the secondary outcome in the two study arms at baseline (baseline screening round).
Baseline cytology (Bethesda classification) | After up to 2 years follow-up
  Number of women with the secondary outcome in the two study arms at baseline (baseline screening round).
Baseline HPV-DNA status | After up to 2 years follow-up
  Prevalence of HPV-infections; HPV-16, -18 and other
Baseline conization | After up to 2 years follow-up
  Number of women with the secondary outcome in the two study arms after baseline screening.

CONTACTS AND LOCATIONS:
Overall Officials: Elsebeth Lynge, Professor, Principal Investigator — University of Copenhagen
Locations (1):
- University of Copenhagen, Copenhagen, Copenhagen K, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ronco G, Dillner J, Elfstrom KM, Tunesi S, Snijders PJ, Arbyn M, Kitchener H, Segnan N, Gilham C, Giorgi-Rossi P, Berkhof J, Peto J, Meijer CJ; International HPV screening working group. Efficacy of HPV-based screening for prevention of invasive cervical cancer: follow-up of four European randomised controlled trials. Lancet. 2014 Feb 8;383(9916):524-32. doi: 10.1016/S0140-6736(13)62218-7. Epub 2013 Nov 3. PMID 24192252
- [Background] Dillner J, Rebolj M, Birembaut P, Petry KU, Szarewski A, Munk C, de Sanjose S, Naucler P, Lloveras B, Kjaer S, Cuzick J, van Ballegooijen M, Clavel C, Iftner T; Joint European Cohort Study. Long term predictive values of cytology and human papillomavirus testing in cervical cancer screening: joint European cohort study. BMJ. 2008 Oct 13;337:a1754. doi: 10.1136/bmj.a1754. PMID 18852164
- [Derived] Thamsborg LH, Andersen B, Larsen LG, Christensen J, Johansen T, Hariri J, Christiansen S, Rygaard C, Lynge E. Danish method study on cervical screening in women offered HPV vaccination as girls (Trial23): a study protocol. BMJ Open. 2018 May 26;8(5):e020294. doi: 10.1136/bmjopen-2017-020294. PMID 29804060